CLINICAL TRIAL: NCT05509244
Title: Efficacy of Acetaminophen-ibuprofen Combination on the Postoperative Pain After Laparoscopic Gynecology Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: acetaminophen-ibuprofen
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): acetaminophen 1g iv dripping
  Interventions: Drug: Acetaminophen
- experimental group (Experimental): the combination of acetaminophen 1g and ibuprofen 300mg iv dripping
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen 1g iv dripping at end of surgery
Drug: Ibuprofen — ibuprofen 300mg iv dripping at end of surgery
  Arms: experimental group

SUMMARY:
Acetaminophen and ibuprofen has been safely used for a long time and reduces postoperative pain and opioid dosages. Investigators are planning to compare the efficacy of 1) acetaminophen only and 2) acetaminophen and ibuprofen combination at postoperative pain after laparoscopic gynecologic surgery.

DETAILED DESCRIPTION:
Acetaminophen and ibuprofen has been safely used for a long time and reduces postoperative pain and opioid dosages. Investigators are planning to compare the efficacy of 1) acetaminophen 1g only and 2) the combination of acetaminophen 1g and ibuprofen 300mg at postoperative pain after laparoscopic gynecologic surgery. Some recovery valuables such as the postoperative pain and opioid requirements will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled gynecologic laparoscopic surgery

Exclusion Criteria:

1. Refusal to be enrolled in the study
2. Emergency surgery
3. On chronic pain medications
4. Psychiatric disorders
5. Pregnant, lactating women
6. Allergy or contraindication to the medication drugs

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-08-24 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | during 30 minutes after surgery
  the maximal postoperative pain severity using pain scale (0=no pain; 10=the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: youngeun moon, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No